CLINICAL TRIAL: NCT00619372
Title: Administration of Anti-CD3 (OKT3) in Combination With Beta-D-Glucosylceramide
Brief Title: Oral OKT3 in Combination With Beta-D-Glucosylceramide
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Ehud Zigmond, M.D., Hadassah University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YI002-HMO-CTIL; Protocol No. 01-300
Record Dates: First submitted 2008-02-10; First posted 2008-02-21 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
Keywords: OKT3; beta-glucosylceramide; oral tolerance; anti-CD3; Safety assessment and healthy volunteers
MeSH Terms: interventions — Muromonab-CD3; Glucosylceramides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- B (Experimental): Low dose OKT3 with GC
  Interventions: Drug: OKT3, GC
- C (Experimental): Mid dose OKT3
  Interventions: Drug: OKT3
- D (Experimental): Mid OKT3 dose with GC
  Interventions: Drug: OKT3, GC
- E (Experimental): High dose OKT3
  Interventions: Drug: OKT3
- F (Experimental): GC only
  Interventions: Drug: GC
- A (Experimental): Low dose OKT3
  Interventions: Drug: OKT3

INTERVENTIONS:
Drug: OKT3 — 0.2 mg OKT3, PO (in the mouth) on day 1 through 5.
  Other Names: OKT3, Monoclonal anti CD3.
  Arms: A
Drug: OKT3, GC — 0.2 mg OKT3 and 7.5 mg GC, PO (in the mouth) on day 1 through 5
  Other Names: OKT3, antiCD3; GC, glucosylceramide, beta glucosylceramide
  Arms: B
Drug: OKT3 — 1 mg OKT3, PO (in the mouth) on day 1 through 5
  Other Names: OKT3, antiCD3
  Arms: C
Drug: OKT3, GC — 1 mg OKT3 and 7.5 mg GC, PO (in the mouth) on day 1 through 5
  Other Names: OKT3, antiCD3; GC, glucosylceramide, beta glucosylceramide
  Arms: D
Drug: OKT3 — 5 mg OKT3, PO (in the mouth) on day 1 through 5
  Other Names: OKT3, anti-CD3; GC, glucosylceramide, beta-glucosylceramide
  Arms: E
Drug: GC — 7.5 mg GC, PO (in the mouth) on day 1 through 5
  Other Names: GC, glucosylceramide, beta glucosylceramide
  Arms: F

SUMMARY:
This clinical study is designed to evaluate the safety of oral administration of the study drug anti CD3 (OKT3) in combination with β-D glucosylceramide [GC] .

DETAILED DESCRIPTION:
Anti CD3 (OKT3): Is an approved drug for intravenous use in the treatment of solid organ transplantation. Preliminary data suggest that the oral administration of OKT3 in low dosages can exert an immune modulatory effect via activation of regulatory T lymphocytes.

β-D glucosylceramide [GC]: Is approved for oral administration and is currently being tested in three clinical trials. Recent data suggested that it can serve as an immunological adjuvant in various clinical settings and to augment the immune response via activation of regulatory T cells.

This clinical trial has been designed to assess the safety of oral administration of OKT3 with and without co-administration of GC in healthy subjects. The use of two potential activators of regulatory T cells, may exert an additive effect, augmenting the systemic immune modulatory effect.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the informed consent process culminating with written informed consent by the subject.
* Men and women > 18 years of age.

Exclusion Criteria:

* Subjects who have undergone surgery within the last 3 months.
* Subjects who have had a prior colostomy, ileostomy, or colectomy with ileorectal anastamosis.
* Subjects presenting with, or who have a history of, persistent intestinal obstruction, bowel perforation, uncontrolled bleeding or abdominal abscess or infection, toxic megacolon.
* Subjects with a clinically significant infectious, immune mediated or malignant disease
* Subjects who are receiving an elemental diet or parenteral nutrition.
* Subjects who have been treated with any time of immune modulatory drug including steroids or NSAID within the last 4 weeks.
* Subjects who have received either methotrexate or cyclosporine or anti TNF alpha (infliximab, Remicade), anti-integrin (namixilab) or who have participated in any other clinical trial within the last 3 months.
* Subjects with a history of coagulopathy.
* Women with childbearing potential unless surgically sterile or using adequate contraception (either IUD, oral or Depo -provera contraceptive, or barrier plus spermicide); pregnant or breastfeeding mothers.
* Subjects who will be unavailable for the duration of the trial, are likely to be non¬compliant with the protocol, or who are felt to be unsuitable by the investigator for any other reason.
* Subjects who are HIV positive
* Subjects who are HBsAg positive
* Subjects who are HCV positive
* Subjects with active CMV
* Subjects who demonstrate a positive PPD
* Subjects with anemia (Hb <10.5 gm/dl)
* Subjects with thrombocytopenia (platelets <100K/microliter)
* Subjects with lymphopenia (absolute lymphocyte count <0.7)
* Subjects with IgG anti-cardiolipin antibody >16 IU
* Prior exposure to OKT3
* Known sensitivity to any ingredients in the study drug

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of the safety of oral administration of OKT3 with and without GC in healthy volunteers by monitoring the subjects for adverse events and by interpreting the results of the various laboratory tests and the subjects' diaries. | January-April

SECONDARY OUTCOMES:
To evaluate the safety of 5 consecutive doses of oral OKT3 with and with out GC and the dose escalation effect in healthy volunteers. | January-April

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Zigmond, M.D., Principal Investigator — Hadassah University Hospital
Locations (2):
- Center for Neurologic Diseases, Brigham and Women's Hospital, Boston, Massachusetts, United States
- Hadassah University Hospital, Jerusalem, Israel